CLINICAL TRIAL: NCT02795611
Title: Effectiveness of Family Centered Occupational Therapy on Play Skills and Participation of Children With Autism Spectrum Disorder
Brief Title: Family Centered Occupational Therapy on Play Skills and Participation of Children With ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201509008RINC
Record Dates: First submitted 2016-05-22; First posted 2016-06-10 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Autism Spectrum Disorder
Keywords: Family-centered; Autism spectrum disorder; Occupational therapy; Participation; Play
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment group (Experimental): Patients who receive 'family-centered occupational therapy' in our hospital
  Interventions: Behavioral: Family-centered occupational therapy
- Control group 1 (Active Comparator): Patients who receive regular occupational therapy in our hospital
  Interventions: Behavioral: regular occupational therapy
- Control group 2 (Other): Patients who don't receive intervention in our hospital
  Interventions: Other: intervention done outside our hospital

INTERVENTIONS:
Behavioral: Family-centered occupational therapy — Caregivers will be equipped with the skills of guiding children with ASD in play and participation in their daily life.
  Arms: Treatment group
Behavioral: regular occupational therapy — regular occupational therapy
  Arms: Control group 1
Other: intervention done outside our hospital — intervention done outside our hospital
  Arms: Control group 2

SUMMARY:
Play skills and participation of children with Autism Spectrum Disorder (ASD) have been restricted by their core symptoms, resulting in heightened parenting stress and affected family daily life. This research aims to improve play skills and participation of children with ASD through 'family-centered occupational therapy', thereby leading to positive outcome for not only the child but also the whole family.

DETAILED DESCRIPTION:
Play skills and participation of children with Autism Spectrum Disorder (ASD) have been restricted by their core symptoms, resulting in heightened parenting stress and affected family daily life. This research aims to improve play skills and participation of children with ASD through 'family-centered occupational therapy', thereby leading to positive outcome for not only the child but also the whole family.

60 children age 2~6 with ASD will be recruited in our research, and divided into either experimental or control groups according to primary caregivers' (will be referred to as caregivers thereafter) decision whether to receive treatment in our hospital (NTUH) or not. Caregivers' decision is based on the convenience of transportation to NTUH. The children with ASD in the experimental group will receive family-centered occupational therapy three times a week for 6 months. The intervention goals, determined by discussing with caregivers, will often be the most important aspect of play skill and participation of children with ASD, which concern caregivers most. Caregivers will be equipped with the skills of guiding children with ASD in play and participation in their daily life. The outcome assessments will include : (1) The child's developmental skills and the severity of ASD as measured with Psychoeducational Profile, third edition (PEP-3) and Childhood Autism Rating Scale (CARS) respectively, (2) the child's play skill and participation as measured with Goal Attainment Scale (GAS), Vineland Adaptive Behavior Scale-Chinese version (VABS-C) and Revised Knox Preschool Play Scale (RKPPS) respectively, (3) Family related factors as measured with Parenting Stress Index Short Form (PSI/SF), Family Outcomes Survey (FOS), Family Empowerment Scale (FES) and Home Observation for Measurement of the Environment (HOME).

Pre- and post-intervention comparison on the outcome measures within the experimental group, and group comparison on the outcome measures will be conducted to examine the effectiveness of family-centered occupational therapy. Results of the study will provide empirical evidence for evidence-based occupational therapy practice in the field of play skills and participation of children with ASD.

ELIGIBILITY:
Inclusion Criteria:

* patient diagnosed with Autism spectrum disorder
* age 2~6 years old

Exclusion Criteria:

* patient with other disease, like seizure or other systemic disease

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2016-05; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Goal Attainment Scale (GAS) | pre-test before intervention and post-test after 3 months and 6 months of intervention
  GAS is a measure we used to assessed change between three time points ("Change from Baseline and at 3 months and at 6 months").
Revised Knox Preschool Play Scale (RKPPS) | pre-test before intervention and post-test after 6 months of intervention
  RKPPS is a measure we used to assessed change between two time points ("Change from Baseline and at 6 months)
Vineland Adaptive Behavior Scale-Chinese version (VABS-C) | pre-test before intervention and post-test after 6 months of intervention
  VABS-C is a measure we used to assessed change between two time points ("Change from Baseline and at 6 months)

SECONDARY OUTCOMES:
Parenting Stress Index Short Form (PSI/SF) | pre-test and post-test after 6 month
Family Outcomes Survey (FOS) | pre-test and post-test after 6 month
Family Empowerment Scale (FES) | pre-test and post-test after 6 month
Home Observation for Measurement of the Environment (HOME) | pre-test and post-test after 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Hui Tseng, PhD, Study Director — National Taiwan University School of Occupational Therapy
Locations (1):
- National Taiwan University Hospital, Taipei, Zhongzheng, Taiwan

IPD SHARING:
Plan to Share IPD: No